CLINICAL TRIAL: NCT02784301
Title: Evaluation of a Biofeedback Tool to Minimize Procedural Pain and Anxiety in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: British Columbia Children's Hospital (Other)
Responsible Party: Principal Investigator, Theresa Newlove, Head, Department of Psychology, British Columbia Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BBAppP2
Record Dates: First submitted 2016-05-17; First posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Belly breathing with biofeedback app (Experimental)
  Interventions: Device: Belly breathing with biofeedback app
- Standard of Care (No Intervention)
- Belly breathing without biofeedback app (Active Comparator)
  Interventions: Behavioral: Belly breathing without biofeedback app
- Belly breathing + visual distraction (Active Comparator)
  Interventions: Behavioral: Belly breathing + visual distraction

INTERVENTIONS:
Device: Belly breathing with biofeedback app — This intervention consists of learning how to belly breathe using a smartphone biofeedback application that coaches children how to breathe slowly and deeply. The app consists of a cartoon avatar in a hot air balloon that inhales and exhales bubbles. The goal of the biofeedback game is to a) teach a voluntary deep breathing protocol, b) detect compliance to the breathing protocol using the attached audio-based pulse oximeter sensor and c) to raise the hot air balloon in accordance to this compliance in order to motivate the children. Scenery changes as the balloon rises, driven by biofeedback, until it eventually reaches outer space.
  Arms: Belly breathing with biofeedback app
Behavioral: Belly breathing without biofeedback app — This intervention consists of learning how to belly breathe without the biofeedback application prior to the blood collection and continuing with self-directed belly breathing during the procedure itself.
  Arms: Belly breathing without biofeedback app
Behavioral: Belly breathing + visual distraction — This intervention consists of learning how to belly breathe without the application plus receiving visual distraction by watching a cartoon avatar in the hot air balloon rising through space. The avatar will not coach the child to breathe as the visual cues for breathing (words and bubbles) will not be present and the avatar will not rise in response to correct belly breathing. Participants will be instructed to continue with self-directed breathing while also watching the visual distraction during the blood collection procedure.
  Arms: Belly breathing + visual distraction

SUMMARY:
Belly breathing is a popular relaxation technique used to reduce anxiety and pain in children during medical procedures. The investigators have developed a biofeedback game that will help teach children how to belly breathe in an interactive way. Existing studies have shown that biofeedback tools are effective ways to teach relaxation techniques to children. The purpose of this study is to evaluate 1) whether this new biofeedback tool is a more a effective and engaging way to teach belly breathing to children and 2) whether the application is more effective in reducing procedural pain and anxiety compared to standard of care, self-directed belly breathing alone or self-directed belly-breathing combined with visual distraction. The investigators hypothesize that:

1. The smartphone-based biofeedback game for belly breathing will reduce self-reported procedural anxiety and pain in children during a blood collection procedure compared to:

   1. standard of care
   2. belly breathing + standard care procedures
   3. belly breathing with visual components of the application with no coaching or biofeedback distraction.
2. The smartphone-based biofeedback game will increase compliance with belly breathing compared to self-directed breathing.
3. Belly breathing with smartphone-based biofeedback game will be more engaging compared to self-directed belly breathing.

DETAILED DESCRIPTION:
1. Purpose

   The purpose of the present study is to evaluate the clinical efficacy of belly breathing using a smartphone-based biofeedback application to reduce procedural anxiety and pain in children having their blood drawn in the blood collection lab at BC Children's Hospital. This phase of the study will focus on evaluating 1) the efficacy of the application in children ages 5-17 for reducing self--reported pain and anxiety during blood collection and 2) the ability of the application to increase belly breathing compliance and engagement compared to traditional teaching methods.
2. Objectives

   The proposed project aims to answer the following questions:
   1. Will the smartphone-based biofeedback game for belly breathing reduce self-reported procedural anxiety and pain in children during a blood collection procedure compared to a) standard of care b) belly breathing + standard care procedures or c) belly breathing with visual components of the application with no coaching or biofeedback distraction?
   2. Will the smartphone-based biofeedback game increase compliance with belly breathing compared to self-directed belly breathing?
   3. Will belly breathing with the smartphone-based biofeedback game be more engaging compared to self-directed belly breathing?
3. Justification

   Belly breathing, a type of deep diaphragmatic breathing that typically produces a relaxed state, is a popular behavioural intervention used to reduce anxiety in children undergoing medical procedures. Studies have shown that decreased anxiety is not only associated with decreased distress but also with decreased pain and less negative attitudes towards future medical procedures. Biofeedback is a tool that is used to teach children about the connection between mind and body. Very little research currently exists on using biofeedback applications to teach relaxation to children in a clinical setting; however, some evidence suggests that it could be effective. This study will examine the efficacy of using such a tool to teach belly breathing to children in order to reduce procedural anxiety and pain.
4. Research Methods

   To explore the above hypotheses, the study design will employ a randomized control trial design. Expected and experienced self-report anxiety and pain scores in children assigned to the belly breathing biofeedback group will be compared to control group scores. The experimental group will be taught to belly breathe using the biofeedback game application and will be instructed to use it during the blood collection procedure. Control Group 1 will receive standard of care. Control Group 2 will receive belly breathing training without the application and be instructed to continue with self-directed belly breathing during the procedure. Control Group 3 will be taught belly breathing without the application plus receive distraction of watching the cartoon avatar in the hot air balloon rising through space; however, the avatar will not 'coach' the child as the visual cues for breathing (words and bubbles) will not be present and the avatar will not rise in response to correct belly breathing. Belly breathing compliance will be measured using extracted respiratory rates from collected PPG data.

   Two trained volunteers will recruit participants in the waiting room of the main blood collection in BC Children's Hospital. They will approach parents and children and invite them to participate in the study. If the parents and child are interested, they will be given consent and assent forms that they can read return to the volunteers at any time before the procedure should they decide to participate.
5. Data Analysis

Pain Scores: An analysis of covariance will be used to determine whether experimental subjects report significantly less pain during blood collection than the control patients. To determine whether belly breathing with the application will alter the expectation of pain, the sample will be divided into high and low expectations of pain using a median split on pain scores. A 2x3 repeated measures analysis of variance will be carried out comparing high and low expectations groups at Time 1, 2, and 3. Paired t-tests will be carried out on the high and low expectation groups within the experimental and control conditions to determine whether there will be any change in expected pain from Time 1 to Time 2.

In order for a clinically significant difference of 2 out 10 in pain score to be detected (alpha=0.05, power 80%) 70 children will be needed per group. In order to allow for non-compliance and post-study exclusions of children with cardiovascular/respiratory conditions or the use of topical anaesthetics, the investigators will need to recruit approximately 300 children.

Anxiety scores: Changes over time in the four groups will be analyzed by time x group interaction in a repeated analysis of variance. Paired T-Tests will be carried out on each of the four groups to determine whether there is any change in anxiety from Time 1 to Time 2.

A Pearson correlation will be used to investigate the relationship between anxiety scores and pain scores in each of the four groups.

Belly Breathing Compliance: Photoplethysmograph (PPG) data collected during blood collection from the experimental group and Control Groups 2 and 3 will be analyzed using a standard peak detection method. Independent Sample T-tests will be carried out on the amplitude of the RSA. Level of significance will be set at p=0.05.

Engagement Scores: The responses to each question on the Study Completion Questionnaires from the Experimental Group and Control Groups 2 and 3 will be analyzed separately using Independent Sample T-Test. Level of significance will be set at p=0.05. The Bonferroni Correction will be used to adjust for multiple measures.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand basic spoken and written English

Exclusion Criteria:

No participants will be excluded from the study. However, data may be excluded during post-study analysis if a child:

* suffers from a severe cardiovascular or respiratory condition that could significantly affect heart rate or respiratory rate
* is taking medication that could significantly affect heart rate or respiratory rate
* is using a local anesthetic during the blood collection procedure

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Self-reported experienced pain | Immediately following blood collection, on average within one minute of needle removal
  Pain will be assessed using the Color Analog Scale (CAS), which is a tool that contains a gradation of colour and width on a piece of plastic, ranging from white and narrow ('no pain') to wide and red ('the most pain') to represent different levels of pain intensity. The child will be instructed to slide a marker along the scale to indicate the colour and width that represents her/his pain and an evaluator then reads and records the corresponding numeral value scored from 0 to 10 in increments of 0.25 on the reverse side of the scale. The slider is originally positioned in the middle of scale. The CAS has been shown to be appropriate for children ages 5 to 18.
Change in self-reported preprocedural anxiety | Prior to blood collection, on average within one minute of consent form completion and five minutes after initial VAS-A score is recorded
  Preprocedural state anxiety will be assessed using the Visual Analogue Scale of Anxiety (VAS-A), which consists of a 100 mm horizontal line with two end points labelled "no anxiety or fear" and "worst possible anxiety or fear." Anxiety will be measured at two time points, prior to and following intervention. The scale will be scored from 1 to 100 (1mm=1/100) and will be presented in a way that the child cannot see his/her previous ratings.
Change in self-reported expected pain | Prior to blood collection, on average within one minute of consent form completion and five minutes after initial CAS score is recorded
  Pain will be assessed twice prior to blood collection using the CAS: once before the intervention and once after the intervention or approximately five minutes after the first assessment for the non-intervention standard of care group.

SECONDARY OUTCOMES:
Belly breathing compliance | During entire blood collection procedure, beginning within ten seconds of sitting in the collection chair and ending within ten seconds of needle removal
  A pulse oximeter will be used to collect a photoplethysmography (PPG) signal, which measures belly breathing compliance through heart rate monitoring.
Belly breathing engagement | Immediately following blood collection; on average the questionnaire will be administered within one minute of needle removal
  A questionnaire with likert-type questions scored on a scale of 1 to 5 (1=strongly disagree; 5=strongly agree) was developed for this study to measure engagement with belly breathing with the application compared to belly breathing without the application.
Self-reported experienced anxiety | Following blood collection, on average within one minute of needle removal
  Procedural state anxiety will be assessed using the VAS-A. The child will be asked to rate the anxiety he/she experienced while he/she was having his/her blood drawn.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Newlove, Ph.D., Principal Investigator — British Columbia Children's Hospital
Locations (1):
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bringuier S, Dadure C, Raux O, Dubois A, Picot MC, Capdevila X. The perioperative validity of the visual analog anxiety scale in children: a discriminant and useful instrument in routine clinical practice to optimize postoperative pain management. Anesth Analg. 2009 Sep;109(3):737-44. doi: 10.1213/ane.0b013e3181af00e4. PMID 19690240
- [Background] Chiang LC, Ma WF, Huang JL, Tseng LF, Hsueh KC. Effect of relaxation-breathing training on anxiety and asthma signs/symptoms of children with moderate-to-severe asthma: a randomized controlled trial. Int J Nurs Stud. 2009 Aug;46(8):1061-70. doi: 10.1016/j.ijnurstu.2009.01.013. Epub 2009 Feb 26. PMID 19246041
- [Background] Claar RL, Walker LS, Smith CA. The influence of appraisals in understanding children's experiences with medical procedures. J Pediatr Psychol. 2002 Oct-Nov;27(7):553-63. doi: 10.1093/jpepsy/27.7.553. PMID 12228327
- [Background] Dehkordi P, Garde A, Karlen W, Wensley D, Ansermino JM, Dumont GA. Pulse rate variability compared with Heart Rate Variability in children with and without sleep disordered breathing. Annu Int Conf IEEE Eng Med Biol Soc. 2013;2013:6563-6. doi: 10.1109/EMBC.2013.6611059. PMID 24111246
- [Background] Elliott CH, Olson RA. The management of children's distress in response to painful medical treatment for burn injuries. Behav Res Ther. 1983;21(6):675-83. doi: 10.1016/0005-7967(83)90086-4. No abstract available. PMID 6661152
- [Background] Huguet A, Stinson JN, McGrath PJ. Measurement of self-reported pain intensity in children and adolescents. J Psychosom Res. 2010 Apr;68(4):329-36. doi: 10.1016/j.jpsychores.2009.06.003. Epub 2009 Oct 2. PMID 20307699
- [Background] Kemper KJ. Complementary and alternative medicine for children: does it work? West J Med. 2001 Apr;174(4):272-6. doi: 10.1136/ewjm.174.4.272. No abstract available. PMID 11290687
- [Background] McDonnell L, Bowden ML. Breathing management: a simple stress and pain reduction strategy for use on a pediatric service. Issues Compr Pediatr Nurs. 1989;12(5):339-44. doi: 10.3109/01460868909038042. PMID 2698873
- [Background] McGrath PA, Seifert CE, Speechley KN, Booth JC, Stitt L, Gibson MC. A new analogue scale for assessing children's pain: an initial validation study. Pain. 1996 Mar;64(3):435-443. doi: 10.1016/0304-3959(95)00171-9. PMID 8783307
- [Background] Powers SW, Mitchell MJ, Byars KC, Bentti AL, LeCates SL, Hershey AD. A pilot study of one-session biofeedback training in pediatric headache. Neurology. 2001 Jan 9;56(1):133. doi: 10.1212/wnl.56.1.133. No abstract available. PMID 11148256
- [Background] Shockey DP, Menzies V, Glick DF, Taylor AG, Boitnott A, Rovnyak V. Preprocedural distress in children with cancer: an intervention using biofeedback and relaxation. J Pediatr Oncol Nurs. 2013 May-Jun;30(3):129-38. doi: 10.1177/1043454213479035. Epub 2013 Mar 29. PMID 23542082
- [Background] Tomlinson D, von Baeyer CL, Stinson JN, Sung L. A systematic review of faces scales for the self-report of pain intensity in children. Pediatrics. 2010 Nov;126(5):e1168-98. doi: 10.1542/peds.2010-1609. Epub 2010 Oct 4. PMID 20921070
- [Background] Tsze DS, von Baeyer CL, Bulloch B, Dayan PS. Validation of self-report pain scales in children. Pediatrics. 2013 Oct;132(4):e971-9. doi: 10.1542/peds.2013-1509. Epub 2013 Sep 2. PMID 23999954
- [Background] Ward CM, Brinkman T, Slifer KJ, Paranjape SM. Using behavioral interventions to assist with routine procedures in children with cystic fibrosis. J Cyst Fibros. 2010 Mar;9(2):150-3. doi: 10.1016/j.jcf.2009.11.008. Epub 2009 Dec 30. PMID 20044315